CLINICAL TRIAL: NCT06327828
Title: Guiding Methimazole Therapy in Graves' Disease - a Randomised Controlled Trial Comparing a Computer-aided Treatment (Digital Thyroid, DigiThy) Versus Usual Care
Brief Title: Methimazole in Graves' Disease - Comparing the Computer-aided Treatment DigiThy Versus Usual Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Graz University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32-663
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-automated computer-aided treatment (Experimental): Treatment based on the dosing suggestions by a mathematical algorithm and cross-checked by the treating physician
  Interventions: Device: Semi-automated computer-aided treatment (Digital Thyroid, DigiThy)
- Usual care (Active Comparator): Treatment based on the dosing suggestions by the treating physician
  Interventions: Procedure: Usual care

INTERVENTIONS:
Device: Semi-automated computer-aided treatment (Digital Thyroid, DigiThy) — Semi-automated computer-aided treatment based on a mathematical model
  Arms: Semi-automated computer-aided treatment
Procedure: Usual care — Guiding methimazole therapy based on the treating physician's decision
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to compare two methods of guiding methimazole therapy in patients with Graves' disease: methimazole dose adjustments based on a new semi-automated computer-guided treatment (based on a mathematical model) or based on the treating physician's decision (i.e. usual care). The main question it aims to answer is whether semi-automated computer-guided treatment is not inferior to usual care in terms of safety, the time it takes to achieve euthyroidism and the methimazole dose required.

ELIGIBILITY:
Inclusion Criteria:

* Active Graves' hyperthyroidism [Thyroid-stimulating hormone <0.1 mU/L, elevated free thyroxine levels (fT4) above the upper limit of normal and positive Thyrotropin receptor antibody (TRAb) according to local laboratory results], measured within the last month prior to the inclusion date
* Patients not yet receiving antithyroid treatment, or having received antithyroid treatment continuously for less than 4 weeks, or relapse or recurrence of Graves' hyperthyroidism defined as patients previously having received and discontinued treatment with antithyroid drugs for at least 4 weeks)
* Age 18 years or older
* Provision of written informed consent

Exclusion Criteria:

* Previous treatment with radioactive iodine
* Ongoing antithyroid treatment for more than one month
* Pregnancy
* Treatment with propylthiouracil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary aim is to compare semi-automated computer-guided treatment with usual care in terms of their performance indices | 18 months
  The performance index is the deviation from the desired free thyroxine (fT4) value

SECONDARY OUTCOMES:
Comparison in terms of cumulative methimazole dosing | 18 months
  Comparison in terms of cumulative methimazole dosing
Comparison based on free thyroxine (fT4) target range | 18 months
  Comparison based on free thyroxine (fT4) target range

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Pilz, MD, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No